CLINICAL TRIAL: NCT01731314
Title: The Learning and Memory of the Experience of Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, MS, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2012P002386
Record Dates: First submitted 2012-11-16; First posted 2012-11-21 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Learning and Memory of Pain

SUMMARY:
This study investigates the learning and memory of pain.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female healthy volunteers.
2. 18-65 years of age.
3. Right-handed.
4. Fluency in English. Ability to read and understand English; English can be a second language provided that the participant feels that he/she is able to understand all the questions used in the assessment measures.

Exclusion Criteria:

1. Any previous experience with conditioned analgesia/hyperalgesia paradigms.
2. Presence of any illness or medication use that is judged to interfere with the trial. For example: psychiatric disorder according to the DSM-IV manual, medication that can influence cognition or emotional processing, i.e. sleep medication, antidepressants, anti-convulsants or opioids.
3. Unwillingness to receive brief pain stimulation administered by a heat probe on the hand.
4. Instability of responses to experimental heat pain
5. Any contraindications to fMRI scanning for subjects in Experiment 2 (including metal implants, claustrophobia, history of head trauma, and pregnancy).
6. Peripheral neuropathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MGH East Campus, 149 13th St., Charlestown, Massachusetts, United States